CLINICAL TRIAL: NCT04960553
Title: Prospective, Open, Non-comparative, Multi-centre, Post Market Clinical Follow-up Investigation to Follow the Progress of Exuding Chronic Wounds to Healing Using Exufiber® as Primary Dressing, and Mepilex® Border Flex/Comfort
Brief Title: A PMCF Investigation on Exuding Chronic Wounds Using Exufiber® as Primary Dressing, and Mepilex® Border Flex/Comfort
Acronym: ExuFlex01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was early terminated because new data related to the investigational device were available making this investigation no longer scientifically relevant
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-708370
Record Dates: First submitted 2021-06-21; First posted 2021-07-14 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Wound Heal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device : Post Market Clinical Follow-up Investigation applying Exufiber® and Mepilex® Border Flex (Experimental): Post Market Clinical Follow-up investigation : Up to 102 subjects with exuding chronic wounds deemed adequate by the Principle Investigator and Clinical Team for assigned treatment
  Interventions: Device: Exufiber® and Mepilex® Border Flex

INTERVENTIONS:
Device: Exufiber® and Mepilex® Border Flex — Post Market Clinical Follow-up Investigation applying Exufiber® and Mepilex® Border Flex to 102 subjects who meet the study criteria for up to 12 weeks

SUMMARY:
The overall objective of this post market clinical follow-up (PMCF) investigation is to follow the progress of exuding chronic wounds to healing, or up to 12 weeks, whichever occurs first, consecutively using Exufiber® as primary dressing, and Mepilex® Border Flex (Mepilex Border Comfort) as primary dressing.

DETAILED DESCRIPTION:
This investigation is as a prospective, open, non-comparative, multi-centre investigation with the aim to follow exuding chronic wound progression. The investigation will include subjects from three populations suffering from exuding chronic wounds (Venous Leg Ulcers, Diabetic Foot Ulcers and Pressure Ulcers). The target wound for all subjects will initially be treated with Exufiber® as primary dressing. As the wound progress and wound exudate production is reduced, the Exufiber will be replaced by the Mepilex Border Flex dressing. For ulcers located at sacrum or heel, the Mepilex Border Heel or Mepilex Border Sacrum will be used.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Both genders ≥18 years old.
* Exuding pressure ulcer, exuding diabetic foot ulcer or exuding venous leg ulcer (an exuding wound defined as one that requires highly absorbent dressing - as per clinical judgement)
* Chronic wound at least 4 weeks duration (chronic would be defined after 4 weeks).
* ABPI (within the last 3 months) ≥0.7 for both legs (if both present). If ABPI >1.4, then big toe pressure >60mmHg is required or an alternative measurement verifying normal distal arterial flow.
* At entry into the study, the ulcer or wound area should be 0.8 cm² - 70 cm².

Exclusion Criteria:

* Known allergy/hypersensitivity to the dressing or its components.
* Subject included in other ongoing clinical investigation at present or during the past 30 days
* Pregnancy or lactation at time of study participation.
* Target wound DFU <0.8 cm² , VLU <3 cm² , PU <1 cm² , post debridement (measured as greatest length x greatest width)
* Infected ulcer according to the judgment of the investigator defined as any wound condition requiring the prescription or continuation of systemic antibiotic therapy at recruitment.
* Other wounds within 3 cm from target wound
* Subject not suitable for the investigation according to the investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Wound progress measured by investigator evaluation | Up to 12 weeks
  Wound progress of exuding chronic wounds from baseline to last visit where Exufiber is applicable, up to 12 weeks.

SECONDARY OUTCOMES:
Wound progress measured by investigator evaluation | Up to 12 weeks
  Wound progress of exuding chronic wounds from baseline to final visit and from first visit where Mepilex Border Flex is applicable as primary dressing to final visit.
Absolute and percentage change in wound area of exuding chronic wounds captured by an independent evaluator evaluating wound photos through the software program PictZar® Digital Planimetry | Up to 12 weeks
  Absolute and percentage change in wound area of exuding chronic wounds, from baseline to last visit where Exufiber is applicable and to final visit; and from first visit where Mepilex Border Flex is applicable as primary dressing to final visit.
Change in necrotic/sloughy tissue of exuding chronic wounds captured through visual judgement by investigator/designee through a scale in percentage | Up to 12 weeks
  Change in necrotic/sloughy tissue of exuding chronic wounds from baseline to last visit where Exufiber is applicable and to final visit; and from first visit where Mepilex Border Flex is applicable as primary dressing to final visit.
Change in granulation tissue of exuding chronic wounds captured through visual judgement by investigator/designee through a scale in percentage | Up to12 weeks
  Assessment of exuding wound from baseline to last visit where Exufiber is applicable and to final visit; and from first visit where Mepilex Border Flex is applicable as primary dressing to final visit.
Changes in peri-wound skin condition of exuding chronic wounds | Up to12 weeks
  Changes in peri-wound skin condition of exuding chronic wounds from baseline to last visit where Exufiber is applicable and to final visit; and from first visit where Mepilex Border Flex is applicable as primary dressing to final visit.
Device usability, wound fluid retention and dressing properties | Up to 12 weeks
  Investigator's evaluation of the wound status and the Exufiber and Mepilex Border Flex dressings, including usability, wound fluid retention and dressing properties.
Subject's perception of pain and comfort | Up to12 weeks
  Subject's perception of Pain and Pain intensity with a numerical rating scale (NRS) range 0-10 cm where 0 is no pain and 10 pain as intense you can imagine. Comfort during Exufiber and Mepilex Border Flex dressings application, removal and use evaluated through questions asked by the investigator/designee to the subject with a range from very poor to very good.
Dressing wear time | Up to12 weeks
  Dressing wear time of the Exufiber dressing and the Mepilex Border Flex dressing, and supporting techniques applied.
Cost-effectiveness | Up to12 weeks
  Cost-effectiveness; wound care consumables and frequency of dressings changes.

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis, Aalst
  - UZ Brussel, Jette
- Portugal (2):
  - Unidade de Cuidados Continuados Ordem da Trindade, Porto
  - Unidade Cuidados Continuados - Mutivaze - WeCare, Póvoa de Varzim
- United Kingdom (3):
  - Northumbria Healthcare NHS Foundation Trust, Ashington
  - Manchester University NHS Foundation Trust, Manchester
  - Salford Royal NHS Foundation Trust, Salford